CLINICAL TRIAL: NCT05598879
Title: Global Cardio Oncology Registry
Acronym: G-COR
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Sadler,Diego, MD FACC Associate Professor of Medicine. CCLCM CWRU, The Cleveland Clinic
Other Study IDs: IRB 22-211
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Hematologic Malignancy; Immune Checkpoint Inhibitor-Related Myocarditis; Cardiotoxicity; Cardiovascular Diseases
Keywords: cardiotoxicity; Cancer related cardiovascular diseases; prospective registry; international collaboration; social determinants of health; health care disparities; real world data; cardiology-oncology team work
MeSH Terms: conditions — Breast Neoplasms; Hematologic Neoplasms; Cardiotoxicity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Breast cancer: Patients with breast cancer who present for initial cardio-oncology consultation. Clinical follow up for 18 months.
  Interventions: Other: anonymized data collection during programmed surveillance clinical follow up
- Hematological malignancies: Patients with lymphomas, leukemias, multiple myeloma, and AL amyloidosis who present for initial cardio-oncology consultation. Clinical follow up for 18 months.
  Interventions: Other: anonymized data collection during programmed surveillance clinical follow up
- Immune check point inhibitors: Patients with any type of cancer treated with immune check point inhibitors who present for initial cardio-oncology consultation. Clinical follow for 18 months
  Interventions: Other: anonymized data collection during programmed surveillance clinical follow up

INTERVENTIONS:
Other: anonymized data collection during programmed surveillance clinical follow up — anonymized data entry of demographic, clinical, imaging, laboratory, cancer treatment, and cardiovascular events into a RedCap Cloud platform

SUMMARY:
G-COR is the first Global Prospective Cardio-Oncology Registry. It is a multinational, multicenter prospective observational cohort registry, with the goal of collecting clinical, laboratory, imaging, demographic, and socioeconomic data to identify risk factors associated with increased incidence of cancer therapy related cardiovascular toxicity (CTR-CVT) in different settings and to derive and validate risk scores for cardio oncology patients treated in different geographic locations throughout the world.

DETAILED DESCRIPTION:
G-COR is the first Global Prospective Cardio-Oncology Registry. It is a multinational, multicenter prospective observational cohort registry, with the goal of collecting clinical, laboratory, imaging, demographic, and socioeconomic data to identify risk factors associated with increased incidence of cancer therapy related cardiovascular toxicity (CTR-CVT) in different settings and to derive and validate risk scores for cardio oncology patients treated in different geographic locations throughout the world.

G-COR will involve the collaboration from 124 hospitals from 24 countries that completed survey with sites demographics. It will evaluate cardiovascular disease in three distinct populations of cancer patients (hematological malignancies: lymphomas, leukemias, multiple myeloma; breast cancer patients; and patients treated with check point inhibitors immunotherapy).

G-COR will evaluate the cardiovascular impact of different cancer treatments in the above-described patients, and similarities and differences in diagnostic and treatment modalities as well as outcomes and the impact of socioeconomic factors and risk factors for toxicities in a large worldwide population.

G-COR will study the impact of cancer in CV disease in cancer patients treated at academic centers as well as in patients treated at community hospitals, through a systematic prospective data collection in a global digital platform.

G-COR is an IRB approved prospective registry, conducted with the logistical support of C5 Clinical Research Division and the Cardiovascular Outcomes Registries and Research (CORR) group at the Cleveland Clinic and have developed eCRFs with an extensive Red Cap Cloud platform.

G-COR Executive, Scientific and topic committees are led by North American, European, Latin American, Australian and Asian representatives from both academic and community centers.

The pilot phase of G-COR enrolls breast cancer patients only, and the global phase will include all three cohorts of patients (breast, Hem and ICIs).

The investigators have started enrolling patients for G-COR pilot phase with US centers, and will start the global international phase in 2023.

ELIGIBILITY:
Inclusion Criteria:

* New cardio-oncology consultation for breast cancer patients, or
* New cardio-oncology consultation for Hodgkin's or non-Hodgkin's lymphoma patients, or
* New cardio-oncology consultation for acute or chronic leukemia patients, or
* New cardio-oncology consultation for multiple myeloma or AL amyloidosis, or
* New cardio-oncology consultations for immune check-point inhibitors cardiac evaluation.
* All patients have to be 18 years old or older

Exclusion Criteria:

* Cardio-oncology patients who have previously had cardio-oncology evaluation and follow up by the investigators.
* Minors less than 18 years old.
* Inability or unwillingness to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity | 18 months of prospective follow up
  Any new cardiac event occurring during or after cancer treatment
New cardiovascular events | 18 months of prospective follow up
  Heart failure, myocardial infarction, cardiac arrhythmias, syncope, coronary revascularization, heart transplant, cerebrovascular accident, peripheral arterial disease, hypertension, pulmonary hypertension. All events will be adjudicated according to standard clinical definitions.
Cardiovascular death. | 18 months of prospective follow up
  Death during or after cancer treatment, adjudicated to cardiovascular causes by treating physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Sadler, MD FACC, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
To be established by the Scientific committee